CLINICAL TRIAL: NCT05878951
Title: A Multicenter Randomized Controlled Trial Examining the Effects of Intra-detrusor Botulinum Toxin at Time of Holmium Laser Enucleation of the Prostate (HoLEP) in Men With Overactive Bladder (OAB) Symptoms
Brief Title: Examining the Effects of Intra-detrusor Botox at Time of HoLEP in Men With Overactive Bladder Symptoms
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Calgary (Other); Ohio State University (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Professor of Urology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00218130
Record Dates: First submitted 2023-05-04; First posted 2023-05-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-07

CONDITIONS: Urinary Incontinence; Overactive Bladder Syndrome; Overactive Bladder; Urologic Diseases
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Urologic Diseases | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intra-detrusor OnabotulinumtoxinA Injection (Experimental): Injection of intra-detrusor OnabotulinumtoxinA into the bladder will be performed.
  Interventions: Drug: OnabotulinumtoxinA
- No intra-detrusor OnabotulinumtoxinA Injection (No Intervention): Injection of intra-detrusor OnabotulinumtoxinA into the bladder will not be performed.

INTERVENTIONS:
Drug: OnabotulinumtoxinA — Intra-detrusor OnabotulinumtoxinA is commonly known as botox
  Other Names: Botox
  Arms: Intra-detrusor OnabotulinumtoxinA Injection

SUMMARY:
The objective of our multi-center randomized single-blind study is to examine the safety and effect of intra-detrusor OnabotulinumtoxinA injections at the time of holium laser enucleation of the prostate (HoLEP) in men with overactive bladder symptoms with and without urge incontinence.

DETAILED DESCRIPTION:
Patients with significant preoperative urgency and/or urge urinary incontinence (UUI) along with lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH) may require post-HoLEP anticholinergic, B-3 agonist, or intravesical OnabotulinumtoxinA administration. This injection is a guideline recommended for treatment in patients with severe irritative LUTS (urgency, UUI) and overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 -89 undergoing HoLEP
* Component of OAB symptoms including frequency, nocturia, urgency, and/or urge related incontinence
* Willing to sign the Informed Consent Form
* Able to read, understand, and complete patient questionnaires.

Exclusion Criteria:

* Allergy or hypersensitivity to OnabotulinumtoxinA injections
* Patients having a concurrent ureteroscopy +/- laser lithotripsy, percutaneous nephrolithotomy, or non-urologic surgery at the time of their HoLEP
* Anticipated need for perineal urethrostomy at the time of HoLEP
* Prior pelvic radiation or patients with a history of bladder cancer with or without BCG therapy
* Patients who lack decisional capacity
* Active urinary tract infection

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men experiencing overactive bladder symptoms
Enrollment: 80 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
Improve Overactive Bladder Symptoms (OAB) utilizing botox injections into the bladder. | 12 months
  Examine the safety and effect of intra-detrusor botulinum toxin injections at the time of helium laser enucleation of the prostate (HoLEP) in men with overactive bladder symptoms with and without urge incontinence.

SECONDARY OUTCOMES:
Difference in safety/ adverse effects | 90 days
  Identifying changes in post-op urinary retention, gross hematuria, UTI, ED visits and any additional complications.
Difference in patient REDCap surveys (gross hematuria dysuria, incontinence) | 6 months
  Identifying symptom resolution at different time points (1 month, 3 months, 6 months)
Difference in efficacy endpoints (3-month clinic/telephone follow-up) | 3 months
  Identifying efficacy endpoints as they relate to the use of anti-cholinergics, incontinence survey, post void residuals, continence pads requirements if any.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Krambeck, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States